CLINICAL TRIAL: NCT02337530
Title: A Randomized Phase II Trial of Selumetinib in Patients Receiving Standard Pemetrexed and Platinum-based Chemotherapy for the Treatment of Advanced or Metastatic KRAS Wildtype or Unknown Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Selumetinib in Patients Receiving Pemetrexed and Platinum-based Chemotherapy in Advanced or Metastatic KRAS Wildtype or Unknown Non-Squamous NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I219
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — AZD 6244; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): Selumetinib: 75mg/ bid PO given on days 2-19 Pemetrexed: 500mg/m^2 & Cisplatin or Carboplatin*: AUC6: 75mg/m^2 given on day 1 Schedule = q 21 days
  *Must be specified at time of randomization. Patients who start on treatment with cisplatin may switch to carboplatin only after discussion with CCTG
  Interventions: Drug: Selumetinib; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Arm B (Active Comparator): Selumetinib: 75mg/ bid PO given on days 1-21 (continuous) Pemetrexed: 500mg/m^2 & Cisplatin*: 75mg/m^2 or carboplatin AUC 6 given on day 1 Schedule = q 21 days
  **Must be specified at time of randomization. Patients who start on treatment with cisplatin may switch to carboplatin only after discussion with CCTG
  Interventions: Drug: Selumetinib; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Arm C (Active Comparator): Selumetinib: NOT GIVEN Pemetrexed: 500mg/m^2 & Cisplatin*: 75mg/m^2 or carboplatin AUC6 given on day 1 Schedule = q 21 days
  *Must be specified at time of randomization. Patients who start on treatment with cisplatin may switch to carboplatin only after discussion with CCTG
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Selumetinib
  Arms: Arm A; Arm B
Drug: Pemetrexed
Drug: Cisplatin
Drug: Carboplatin

SUMMARY:
The purpose of this study is to find out what effects a new drug, selumetinib, has on lung cancer when receiving standard chemotherapy with pemetrexed and platinum-based chemotherapy.

DETAILED DESCRIPTION:
This research is being done to see whether selumetinib improves the results of standard chemotherapy. The standard or usual treatment for this disease is treatment with chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and/or cytologically confirmed non-squamous, KRAS wildtype or unknown, non-small cell lung cancer that is stage IIIB or IV, metastatic or unresectable and for which standard curative measures do not exist.
* All patients must have a formalin fixed paraffin embedded tumour block (from primary or metastatic tumour) available for correlative studies and must have provided informed consent for the release of the block for correlative studies.
* Patients must have at least one site of disease which is unidimensionally measurable as follows:
* Measurable disease defined as at least one target lesion that has not been irradiated or has progressed after radiation and can be accurately measured in at least one dimension by RECIST 1.1 criteria.
* Chest X-ray ≥ 20 mm
* CT/MRI scan (with slice thickness of < 5 mm) ≥ 10 mm --> longest diameter
* Physical exam (using calipers) ≥ 10 mm
* Lymph nodes by CT scan ≥ 15 mm --> measured in short axis
* Presence of clinically and/or radiologically documented disease (marker positive only patients are not eligible). All radiology studies must be performed within 28 days prior to randomization (within 35 days if negative).
* Age ≥ 18 years.
* ECOG performance status 0 or 1
* Previous Therapy Surgery: Previous major surgery is permitted provided it has been at least 14 days prior to patient randomization and that wound healing has occurred.

Radiation: Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and enrollment to the trial.

Chemotherapy and systemic therapy: Prior therapy with ALK inhibitors is permissible. Patients may not have received prior MEK inhibitors or any other tyrosine kinase inhibitor (including EGFR inhibitors of any kind). Patients may have received vaccines, immunotherapy or other agents that are not MEK/tyrosine kinase inhibitors in the adjuvant setting or for advanced or metastatic disease.

Prior adjuvant platinum-based chemotherapy or combined chemoradiotherapy with curative intent is permissible provided completed at least one year prior to enrollment. No prior cytotoxic chemotherapy for advanced / metastatic disease is permissible.

- Laboratory Requirements (must be done within 7 days prior to randomization)

Neutrophils ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L

Biochemistry:

Creatinine Clearance* ≥ 50 ml/min Total bilirubin ≤ 1.5 x ULN AST and ALT ≤ 2.5 x ULN (if liver metastases ≤ 5x UNL permissible providing ALP also ≤ 6 x UNL)

* Creatinine clearance to be measured directly by 24 hour urine sampling or as calculated by appropriate formula below: Females: GFR = 1.04 x (140-age) x weight in kg/serum creatinine in μmol/L Males: GFR = 1.23 x (140-age) x weight in kg/serum creatinine in μmol/L

* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate
* Patients must be accessible for treatment and follow-up. Patients randomized on this trial must be treated and followed at the participating centre
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient randomization

Exclusion Criteria:

* Patients with a history of other untreated malignancies or malignancies which required therapy within the past 2 years
* No symptomatic brain metastases or spinal cord compression. Patients with asymptomatic brain/spinal cord metastasis who are not planned for radiation, or who have been treated and are stable off steroids (or on a decreasing dose) and anticonvulsants are eligible.
* Patients with significant cardiac disease, including:
* any factors that increase the risk of QTc prolongation or risk of arrhythmic events (e.g. heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age) or mean resting corrected QT interval (QTc) > 470 msec
* uncontrolled hypertension (BP ≥ 150/95 mmHg despite medical therapy)
* acute coronary syndrome within 6 months prior to starting treatment
* angina Canadian Cardiovascular Society Grade II-IV (despite medical therapy)
* symptomatic heart failure (NYHA II-IV)
* prior or current cardiomyopathy
* atrial fibrillation with a ventricular rate > 100 bpm at rest
* severe valvular heart disease Patients with cardiac disease, who do not meet the exclusion criteria above, must have a baseline LVEF ≥ 50%.
* Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
* Patients who have neuropathy > grade 1 or other conditions precluding treatment with the standard chemotherapy regimen planned. Consult CCTG for patients with localised neuropathies as such patients may be eligible.
* Patients who have significant gastrointestinal disease and who are unable to swallow capsules.
* Patients on potent inhibitors or inducers of CYP3A4/5, CYP2C19 and CYP1A2 (must have discontinued within 2 weeks prior to randomization or 3 weeks for St. John's Wort). Patients who do not agree to avoid the ingestion of large amounts of grapefruit and Seville oranges (and other products containing these fruits, e.g. grapefruit juice or marmalade) and not take vitamin E supplements or multivitamin supplements.

Patients who require oral anticoagulants (Coumadin) are eligible provided there is increased vigilance with respect to INR monitoring upon initiation of dosing with selumetinib. If medically appropriate and treatment available, the investigator should consider switching these patients to LMW heparin.

* Patients with current or past history of central serous retinopathy or retinal vein occlusion, high intraocular pressure (≥ 21mm) or uncontrolled glaucoma (irrespective of IOP). Patients with visual symptoms should undergo ophthalmologic examination prior to randomization.
* Pregnant or lactating women. Women of childbearing potential must have a urine pregnancy test proven negative within 7 days prior to randomization. Men and women of childbearing potential must agree to use adequate contraception
* Patients who do not agree to avoid excessive sun exposure and use adequate sunscreen protection.
* Selumetinib-specific precautions for patients of Asian ethnicity:

Plasma exposure of selumetinib (Cmax and AUC) is higher, at a population level, in subjects of Asian descent by approximately 1.5- to 2-fold in non-Japanese Asians and Japanese subjects, compared with Western subjects. However, there is overlap in the range of exposure experienced by Asian and Western subjects and the higher average plasma exposure was not associated with a change in the tolerability profile of single dose selumetinib.

Investigators should make a clinical judgment as to whether the potential risk of experiencing higher selumetinib plasma exposure and potential adverse events outweighs the potential benefit of treatment with selumetinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-05-26 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Penelope A Bradbury, Study Chair — Univ. Health Network-Princess Margaret Hospital, Toronto ON Canada; Barbara Lynn Melosky, Study Chair — BCCA - Vancouver Cancer Centre, Vancouver BC Canada
Locations (12):
- Canada (12):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Abbotsford Centre, Abbotsford, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - Regional Health Authority B, Zone 2, Saint John, New Brunswick
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Melosky B, Bradbury P, Tu D, Florescu M, Reiman A, Nicholas G, Basappa N, Rothenstein J, Goffin JR, Laurie SA, Wheatley-Price P, Leighl N, Goss G, Reaume MN, Butts C, Murray N, Card C, Ko J, Blais N, Gray S, Lui H, Brown-Walker P, Kaurah P, Prentice LM, Seymour L. Selumetinib in patients receiving standard pemetrexed and platinum-based chemotherapy for advanced or metastatic KRAS wildtype or unknown non-squamous non-small cell lung cancer: A randomized, multicenter, phase II study. Canadian Cancer Trials Group (CCTG) IND.219. Lung Cancer. 2019 Jul;133:48-55. doi: 10.1016/j.lungcan.2019.04.027. Epub 2019 May 1. PMID 31200828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between February 2015 and May 2017 from cancer centres in Canada.
Groups:
- Intermittent Oral Selumatinib With Pemetrexed and Platinum: Selumetinib: 75mg/ bid PO given on days 2-19 Pemetrexed: 500mg/m^2 & Cisplatin or Carboplatin*: AUC6: 75mg/m^2 given on day 1 Schedule = q 21 days
  *Must be specified at time of randomization. Patients who start on treatment with cisplatin may switch to carboplatin only after discussion with CCTG
  Selumetinib
  Pemetrexed
  Cisplatin
  Carboplatin
- Continuous Oral Selumatinib With Pemetrexed and Platinum: Selumetinib: 75mg/ bid PO given on days 1-21 (continuous) Pemetrexed: 500mg/m^2 & Cisplatin*: 75mg/m^2 or carboplatin AUC 6 given on day 1 Schedule = q 21 days
  **Must be specified at time of randomization. Patients who start on treatment with cisplatin may switch to carboplatin only after discussion with CCTG
  Selumetinib
  Pemetrexed
  Cisplatin
  Carboplatin
- Pemetrexed and Platinum Alone: Selumetinib: NOT GIVEN Pemetrexed: 500mg/m^2 & Cisplatin*: 75mg/m^2 or carboplatin AUC6 given on day 1 Schedule = q 21 days
  *Must be specified at time of randomization. Patients who start on treatment with cisplatin may switch to carboplatin only after discussion with CCTG
  Pemetrexed
  Cisplatin
  Carboplatin
Period: Overall Study
Arm/Group | Intermittent Oral Selumatinib With Pemetrexed and Platinum | Continuous Oral Selumatinib With Pemetrexed and Platinum | Pemetrexed and Platinum Alone
Started | 20 | 21 | 21
Completed | 20 | 21 | 21
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intermittent Oral Selumatinib With Pemetrexed and Platinum | Continuous Oral Selumatinib With Pemetrexed and Platinum | Pemetrexed and Platinum Alone | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 10 | 33
  >=65 years | 9 | 9 | 11 | 29
Age, Continuous [Median (Full Range); unit: years] | 68 [50 to 80] | 66 [53 to 82] | 65 [42 to 85] | 66 [42 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 11 | 32
  Male | 10 | 10 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 21 | 21 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 21 | 21 | 62
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 4 | 3 | 3 | 10
    1 | 16 | 18 | 18 | 52

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Defined as percentage of participants with objective response over all participants randomized. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.
Time Frame: 2 years and 5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intermittent Oral Selumatinib With Pemetrexed and Platinum | Continuous Oral Selumatinib With Pemetrexed and Platinum | Pemetrexed and Platinum Alone
Number analyzed (Participants) | 20 | 21 | 21
Participants
  Responded | 6 | 14 | 5
  Not Responded | 14 | 7 | 16
Statistical Analysis 1: Comparison: Intermittent Oral Selumatinib With Pemetrexed and Platinum vs Pemetrexed and Platinum Alone; Test type: Superiority; p = 0.73, Fisher Exact; Odds Ratio (OR) = 1.37, 95% CI 2-sided [0.28 to 7.01]
Statistical Analysis 2: Comparison: Continuous Oral Selumatinib With Pemetrexed and Platinum vs Pemetrexed and Platinum Alone; Test type: Superiority; p = 0.01, Fisher Exact; Odds Ratio (OR) = 6.40, 95% CI 2-sided [1.65 to 24.8]

2. Secondary Outcome: Progression Free Survival
Description: Defined as the time from randomization to the first objective documentation of disease progression, defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions, or death due to any cause with patients who had not progressed or died at the time of final analysis censored on the date of the last tumour assessment.
Time Frame: 2 years 5 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Intermittent Oral Selumatinib With Pemetrexed and Platinum | Continuous Oral Selumatinib With Pemetrexed and Platinum | Pemetrexed and Platinum Alone
Number analyzed (Participants) | 20 | 21 | 21
months | 7.2 [4.0 to 8.6] | 6.9 [4.6 to 8.6] | 4.0 [1.4 to 6.8]
Statistical Analysis 1: Comparison: Intermittent Oral Selumatinib With Pemetrexed and Platinum vs Continuous Oral Selumatinib With Pemetrexed and Platinum; Test type: Superiority; p = 0.56, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.42 to 1.60]
Statistical Analysis 2: Comparison: Continuous Oral Selumatinib With Pemetrexed and Platinum vs Pemetrexed and Platinum Alone; Test type: Superiority; p = 0.44, Log Rank; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.40 to 1.49]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Intermittent Oral Selumatinib With Pemetrexed and Platinum | Continuous Oral Selumatinib With Pemetrexed and Platinum | Pemetrexed and Platinum Alone
All-Cause Mortality (participants affected / at risk) | 13/20 | 15/21 | 9/21
Serious Adverse Events (participants affected / at risk) | 14/20 | 14/21 | 9/21
Other Adverse Events (participants affected / at risk) | 20/20 | 21/21 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent Oral Selumatinib With Pemetrexed and Platinum (N=20) | Continuous Oral Selumatinib With Pemetrexed and Platinum (N=21) | Pemetrexed and Platinum Alone (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 1
Other eye disorders (Eye disorders) | 1 | 0 | 0
Colonic perforation (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 0
Edema limbs (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 2
Bronchial infection (Infections and infestations) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 2 | 2 | 2
Pleural infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Other neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Stroke (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Delusions (Psychiatric disorders) | 0 | 0 | 1
Hallucinations (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 6 | 1 | 1
Vasculitis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intermittent Oral Selumatinib With Pemetrexed and Platinum (N=20) | Continuous Oral Selumatinib With Pemetrexed and Platinum (N=21) | Pemetrexed and Platinum Alone (N=21)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 4
Tinnitus (Ear and labyrinth disorders) | 2 | 4 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0
Blurred vision (Eye disorders) | 3 | 2 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 2 | 1 | 1
Watering eyes (Eye disorders) | 4 | 3 | 6
Other eye disorders (Eye disorders) | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 3
Bloating (Gastrointestinal disorders) | 4 | 0 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 12 | 15 | 18
Diarrhea (Gastrointestinal disorders) | 11 | 13 | 9
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 5 | 3
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 4 | 2
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 3 | 1 | 2
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 9 | 6
Nausea (Gastrointestinal disorders) | 14 | 16 | 17
Oral hemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Oral pain (Gastrointestinal disorders) | 2 | 1 | 1
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 2 | 0
Vomiting (Gastrointestinal disorders) | 12 | 16 | 13
Other gastrointestinal disorders (Gastrointestinal disorders) | 1 | 2 | 0
Chills (General disorders) | 0 | 2 | 1
Edema face (General disorders) | 4 | 5 | 4
Edema limbs (General disorders) | 11 | 16 | 11
Fatigue (General disorders) | 19 | 20 | 18
Fever (General disorders) | 3 | 2 | 2
Flu like symptoms (General disorders) | 1 | 2 | 1
Localized edema (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 4 | 3 | 5
Pain (General disorders) | 4 | 5 | 4
Other general disorders, administration site conditions (General disorders) | 1 | 0 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 2
Mucosal infection (Infections and infestations) | 3 | 4 | 0
Paronychia (Infections and infestations) | 1 | 1 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin infection (Infections and infestations) | 3 | 4 | 0
Upper respiratory infection (Infections and infestations) | 2 | 2 | 3
Urinary tract infection (Infections and infestations) | 2 | 1 | 1
Other infections and infestations (Infections and infestations) | 2 | 2 | 2
Bruising (Injury, poisoning and procedural complications) | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Weight loss (Investigations) | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 11 | 15 | 11
Dehydration (Metabolism and nutrition disorders) | 4 | 5 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 4 | 2
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 4 | 11
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7 | 5
Dizziness (Nervous system disorders) | 1 | 10 | 5
Dysgeusia (Nervous system disorders) | 2 | 4 | 2
Headache (Nervous system disorders) | 6 | 9 | 7
Memory impairment (Nervous system disorders) | 1 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 4 | 5
Syncope (Nervous system disorders) | 1 | 2 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0
Other nervous system disorders (Nervous system disorders) | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 3 | 3 | 6
Confusion (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 1
Insomnia (Psychiatric disorders) | 9 | 9 | 6
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 3 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 15 | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 16 | 14
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1
Other respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 6 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 4 | 7 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 | 9 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 7 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Other skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 | 3 | 3
Hematoma (Vascular disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 3 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 2
Hypotension (Vascular disorders) | 1 | 5 | 0
Thromboembolic event (Vascular disorders) | 4 | 8 | 5
Visceral arterial ischemia (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT02337530/Prot_SAP_000.pdf